CLINICAL TRIAL: NCT06018480
Title: NADPH Oxidase Affects on Blood Flow After Administering a High Carbohydrate Meal Pre- and Post-creatine Monohydrate Supplementation.
Brief Title: The Effect of NADPH Oxidase and Creatine Supplementation on Microvascular Blood Flow Regulation
Acronym: NOXCROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Paul Baker, Graduate Research Assistant, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003857
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Endothelial Dysfunction
Keywords: Blood Flow; Endothelial Function; Supplementation
MeSH Terms: interventions — Creatine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Monohydrate Supplementation (Experimental): Participants will be provided with 20 grams of creatine monohydrate per day (100 grams total) in sealed and unopened packages (5 grams in each package). Participants will be asked to complete their supplementation protocol (20 grams/day) by mixing 5 grams of creatine monohydrate powder into water 4 times a day or 10 grams of creatine monohydrate powder into water twice a day. This supplementation will occur after a baseline visit in which participants consume a high-carb meal and have their vascular function studied before the meal and four hours post-prandial. Following the 5 days of supplementation participants will come back and consume a high-carb meal and have their vascular function studied before the meal and four hours post-prandial.
  Interventions: Other: Creatine Monohydrate
- Placebo (Maltodextrin) (Placebo Comparator): Participants will be provided with 20 grams of maltodextrin (placebo) per day (100 grams total) in sealed and unopened packages (5 grams in each package). Participants will be asked to complete their supplementation protocol (20 grams/day) by mixing 5 grams of maltodextrin (placebo) into water 4 times a day or 10 grams of maltodextrin (placebo) powder into water twice a day. This supplementation will occur after a baseline visit in which participants consume a high-carb meal and have their vascular function studied before the meal and four hours post-prandial. Following the 5 days of supplementation participants will come back and consume a high-carb meal and have their vascular function studied before the meal and four hours post-prandial.
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Other: Creatine Monohydrate — The supplementation is the intervention.
  Other Names: AlzChem
  Arms: Creatine Monohydrate Supplementation
Other: Maltodextrin (Placebo) — Placebo to Creatine Monohydrate
  Arms: Placebo (Maltodextrin)

SUMMARY:
This research study seeks to determine the effects of an enzyme in the human body called NADPH oxidase (NOX) on blood flow. In addition, the study will investigate the benefits of creatine monohydrate, a common sports performance supplement, on blood food and vessel function. Participants will undergo two study arms, one in which they consume a high carbohydrate meal pre- and post-creatine monohydrate supplementation and one in which they will consume a high carbohydrate meal pre- and post-placebo supplementation. Blood flow and endothelial function will be assessed before and for 4 hours following the consumption of a high-carbohydrate meal pre and post-supplementation (creatine monohydrate and placebo).

DETAILED DESCRIPTION:
A double-blind cross-over placebo-controlled study design will be used to determine the extent to which NOX and creatine monohydrate supplementation influences skeletal muscle microvascular blood flow and endothelial function following the administration of a high carbohydrate meal in sedentary individuals with overweight/obesity. Participants will be initially screened through a telephone screening over the phone or through an electronic copy (Qualtrics survey) and upon meeting the inclusion criteria, will be scheduled for a baseline visit. At the baseline visits participants will go through an informed consent, background and medical history questionnaire alongside a Dual-energy X-ray absorptiometry (DXA) scan and indirect calorimetry. Subsequently, participants will undergo two main testing days, one will occur before supplementation (creatine monohydrate or placebo) and the other following five days of supplementation (creatine monohydrate or placebo). At the main testing days participants will have their resting blood flow and endothelial function assessed before and for 4 hours following the consumption of a high carbohydrate meal. Following the two main testing days in the first study arm, participants will then undergo a 4-week wash-out in which they will resume their normal behavior and stop taking the supplement they were provided. After the washout period, participants will come back and repeat the baseline visit and the two main testing days. The only difference is that participants will receive the other treatment that was not received the first time (creatine monohydrate or placebo). Which treatment the participant receives first or second will be at random.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 25.0-34.9 kg/m2
* Sedentary; sedentary status will be defined as not performing purposeful exercise training more than 20 minutes per day three a week.
* Currently residing in Tallahassee, Florida, or the surrounding area
* Not taking any medication(s) that interfere with metabolism.
* Not taking any antioxidant supplementation, at least four weeks before the study.
* Not supplementing with creatine monohydrate, at least four weeks before the study.
* Not smoking, vaping, or chewing tobacco and willing to refrain from smoking, vaping, and chewing tobacco throughout the entire study.
* Are not pregnant or planning on becoming pregnant

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, and any condition that interferes with metabolism or oxygen delivery/transport including:

  * Diagnosed cardiovascular diseases or previous myocardial infarction.
  * Uncontrolled hypertension (resting: above 140 mmHg systolic or 90 mmHg diastolic)
  * Diabetes (Type 1 or 2)
  * Uncontrolled thyroid conditions
* Cigarette smoking: current cigarette smoker or those who quit within the previous 6 months.
* Participants consuming supplements or medication known to impact metabolism.
* Participants already consuming creatine monohydrate
* Allergies or intolerance to foods included in the standardized and high carbohydrate meal.
* Women that are pregnant or planning on becoming pregnant
* Weight gain or loss > 10% of body weight during the past 6 months
* Participants consume a vegan or vegetarian diet.
* Non-English-speaking individuals, infants, children, teenagers, cognitively impaired adults individuals, and adults who are unable to consent will be recruited for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Concentrations of reactive oxygen species (ROS) | Change from pre to post five days of creatine monohydrate supplementation at 0, 1, 2, 3, 4 hours post high carbohydrate meal
  Reactive oxygen species measured with microdialysis, reported as hydrogen peroxide (H2O2) concentrations.
Rate of skeletal muscle blood flow | Change from pre to post five days of creatine monohydrate supplementation at 0, 1, 2, 3, 4 hours post high carbohydrate meal
  Skeletal muscle microvascular blood flow measured with microdialysis reported as ethanol outflow/inflow ratio which is inversely with blood flow.
Flow mediated dilation percentage | Change from pre to post five days of creatine monohydrate supplementation at 0, 1, 2, 3, 4 hours post high carbohydrate meal
  Endothelial function as measured with brachial artery flow-mediated dilation, reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Baker, MS, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No